CLINICAL TRIAL: NCT04476238
Title: Randomized Cross-over Trial to Investigate the Effect of Inosine on Human Energy Expenditure
Brief Title: Inosine Energy Expenditure Study
Acronym: InoBAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2020-01026
Record Dates: First submitted 2020-07-14; First posted 2020-07-20 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Healthy Volunteers
Keywords: Energy expenditure; metabolism; inosine
MeSH Terms: interventions — Inosine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inosine (Experimental): 2 grams of inosine dissolved in 250 ml of tap water
  Interventions: Dietary Supplement: Inosine
- Water (Placebo Comparator): 250 ml of tap water only
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Inosine — 2 grams of inosine dissolved in 250 ml water taken by mouth
  Arms: Inosine
Other: Placebo — 250 ml water taken by mouth
  Arms: Water

SUMMARY:
Investigators want to test whether the intake of the nucleoside inosine increases the human energy expenditure. Inosine occurs as a metabolic intermediate in the human body and is sometimes taken as a dietary supplement by athletes.

For this purpose, investigators will measure the basal metabolic rate by indirect calorimetry. Study participants will then take inosine dissolved in water or placebo and energy expenditure will be assessed again.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* BMI between 18-27 kg/m2
* Age between 18 and 40 years

Exclusion Criteria:

* Chronic concomitant disease states (e.g., renal failure, hepatic dysfunction, cardiovascular disease, diabetes mellitus),
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the study
* Participation in another study with investigational drug within the 30 days preceding and during the present study,
* Previous enrolment into the current study,
* Enrolment of the investigator, his/her family members, employees and other dependent persons,
* Thyroid disorders

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2022-02-28 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
resting energy expenditure after Inosine | one hour after oral intake of inosine
  resting energy expenditure (REE) assessed by indirect calorimetry after oral intake of two grams of inosine as compared to placebo

SECONDARY OUTCOMES:
Change in energy expenditure | one hour after oral intake of inosine
  - Difference in EE between baseline measurement and measurement one hour after administration of inosine or control, respectively, at each study visit.
Change in Respiratory Quotient | one hour after oral intake of inosine
  - Respiratory quotient (RQ) as an indicator of substrate oxidation one hour after oral intake of two grams of inosine
Serum inosine level | 0 hours, 1 hour, 2 hours
  Serum inosine levels after ingestion of inosine

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Basel, Department of Endocrinology, Basel, Canton of Basel-City, Switzerland

IPD SHARING:
Plan to Share IPD: No